CLINICAL TRIAL: NCT02541955
Title: Use of Acthar in Rheumatoid Arthritis Related Flares
Brief Title: Use of Acthar in Rheumatoid Arthritis (RA) Related Flares
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Veena Ranganath, MD, MS (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor-Investigator, Veena Ranganath, MD, MS, Assistant Clinical Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Acthar in Rheumatoid Arthritis
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid arthritis (RA); Musculoskeletal ultrasound (MSUS)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 40 Units (Active Comparator): 40 units of Acthar per week
  Interventions: Drug: Acthar
- 80 Units (Active Comparator): 80 units of Acthar twice per week
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — Injections will be self administered
  Other Names: Repository corticotropin injection

SUMMARY:
This is a Rheumatoid Arthritis (RA) study. The purpose of this research study is to determine in RA flare, whether musculoskeletal ultrasound (MSUS) inflammatory scores and/or disease activity scores improve with Acthar treatment.

DETAILED DESCRIPTION:
Participants with active RA flair will be assigned to take on one of two Acthar doses, either 40 units per week or 80 units twice a week. Both arms will be taking the drug for 4 weeks. Each participant will be coming back for visits at 2 weeks, 1 month and 3 months after the initial baseline visit. During these visits the following information will be collected: MSUS of joints, DAS28, Clinical Disease Activity Index (CDAI), Routine Assessment of Patient Index Data 3 (RAPID3) and Health Assessment Questionnaire-Disability Index (HAQ-DI). Participants will also be asked to fill out a questionnaire about their health status.

Efficacy of Acthar to decrease evidence of MSUS synovitis and disease activity measures will be analyzed using the above mentioned instruments, as well as Acthar's ability to prevent the necessity to change patients' RA treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must meet 1987 ACR criteria
2. Age > 18 years of age
3. Baseline DAS28/Erythrocyte Sedimentation Rate (ESR) >=3.2
4. Stable concomitant Disease Modifying Anti-Rheumatic Drugs (DMARDs)
5. Stable prednisone <10mg or equivalent
6. Power Doppler score of >=10

Exclusion Criteria:

1. Prior treatment with Acthar in the past 2mos
2. Meet one of the above RA flare requirements
3. Subjects who have received live or live attenuated vaccines within 6 weeks prior to the first dose of study drug (or the zoster vaccine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Ultrasound Power Doppler Score | Baseline to 2 Weeks
  Using Ultrasound a measure of Power Doppler will be calculated. The change in the scores will be analyzed between the two groups.
DAS28 | Baseline to 2 Weeks
  DAS28 will be calculated. The change in the scores will be analyzed between the two groups.

SECONDARY OUTCOMES:
Ultrasound Grey Scale Synovial Hypertrophy score | Baseline to 2 Weeks
  Using Ultrasound a measure of Grey Scale Synovial Hypertrophy will be calculated. The change in the scores will be analyzed between the two groups.
HAQ-DI | Baseline to 4 Weeks
  Self-administered HAQ-DI summary score will be calculated. The change in the scores will be analyzed between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Veena K Ranganath, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States